CLINICAL TRIAL: NCT02614664
Title: Changes in Cerebral Oxygenation During Laparoscopy in Patients With Single Ventricle Anatomy
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator moved to another institution.
Sponsor: Roby Sebastian (Other)
Responsible Party: Sponsor-Investigator, Roby Sebastian, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00821
Record Dates: First submitted 2015-11-13; First posted 2015-11-25 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Congenital Heart Disease; Single Ventricle
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single ventricle: Patients with single ventricle physiology presenting for laparoscopic procedures.
  Interventions: Device: NIRS

INTERVENTIONS:
Device: NIRS — Cerebral oxygenation monitor which is standard of care for this surgery.

SUMMARY:
Patients with single ventricle physiology (hypoplastic left heart syndrome, tricuspid atresia) frequently have feeding difficulties necessitating procedures such as Nissen fundoplication and G-tube placement. With advances in minimally invasive surgery, these are frequently performed using laparoscopic techniques. Although generally safe and effective, the increase in IAP during laparoscopy may increase systemic and pulmonary vascular resistance and decrease cardiac output. This prospective study will include 50 patients with single ventricle physiology presenting for laparoscopic procedures. There will be no change in the anesthetic or perioperative care of these patients. Tissue and cerebral oxygenation will be monitored using near infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with single ventricle physiology presenting for laparoscopic procedures.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with single ventricle anatomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2017-10-11 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Change in cerebral oxygenation values | From baseline to insufflation (average time frame of 30 mins. - 2 hrs.)
  Measured on the NIRS cerebral oxygenation monitor attached to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Roby Sebastian, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No